CLINICAL TRIAL: NCT05509751
Title: Supporting Older Adults With Cancer and Their Support Person Through Geriatric Assessment and Remote Exercise and Education: the SOAR Study
Brief Title: The SOAR Study: a Study of Geriatric Assessment and Exercise for Older Adults and Their Support Person
Acronym: SOAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martine Puts (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Martine Puts, Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTO#4087
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Gastro-intestinal Cancer; Genito-Urinary Cancer; Breast Cancer; Gynecologic Cancer; Lymphoma
Keywords: comprehensive geriatric assessment; chair-based exercise; health education
MeSH Terms: conditions — Lung Neoplasms; Urogenital Neoplasms; Breast Neoplasms; Lymphoma; Health Education | interventions — Exercise; Geriatric Assessment; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study statistician will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Active Comparator): geriatric assessment (GAM) and remote exercise and education prior to and during curative/adjuvant or first/second line palliative chemotherapy /immunotherapy or targeted therapy
  Interventions: Behavioral: GAM, exercise, health education
- Waitlist control group (No Intervention): Wait list, receiving standard of care and option to receive intervention after treatment.
- single arm pre-post test study for participants recruited from geriatric oncology clinic (Experimental): They will receive the 12 week virtual chair-based exercise and health education intervention except no geriatric assessment
  Interventions: Behavioral: online chair-based exercise combined with health education

INTERVENTIONS:
Behavioral: GAM, exercise, health education — geriatric assessment, exercise and health education
  Other Names: Comprehensive Geriatric Assessment and Management (GAM) combined with online chair-based exercise (CBE) and health education for 12 weeks.
  Arms: Intervention group
Behavioral: online chair-based exercise combined with health education — online chair-based exercise and health education for 12 weeks
  Arms: single arm pre-post test study for participants recruited from geriatric oncology clinic

SUMMARY:
Phase 2 randomized controlled study using a waitlist control group. The study also has a single arm pre-post test 12-week chair-based exercise arm for those who have received the geriatric assessment in the older adults with cancer clinic (geriatric oncology clinic).

Study Duration 2.5 years

Study Agent/ Intervention/ Procedure Comprehensive Geriatric Assessment and Management (GAM) combined with online chair-based exercise (CBE) and health education for 12 weeks.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to compare the standard of care alone to using a detailed health assessment for older adults followed by a 12 week program of online physical activity and health education (also called the intervention) plus the standard of care. The addition of the detailed health assessment for older adults followed by a 12 week program of online physical activity and health education to the standard of care could benefit older adults with cancer in terms of improving their physical activity, muscle strength, quality of life, and fatigue.

The intervention group will receive a detailed health assessment for older adults followed by a 12- week program of physical activity and health education. During the assessment they will be asked to provide information on current health, mood, weight loss, vision and hearing, memory, fatigue, pain, and a review of medications. Additionally, they will be asked to undergo a few tests that assess walking, grip strength, and balance and complete questionnaires that evaluate quality of life, fatigue, anxiety, depression, and physical function.

Two weekly sessions of group-based exercise (20-40) minutes are conducted via Zoom by a qualified exercise professional. These sessions include aerobic exercise for 20 minutes; resistance training, for 10 minutes; balance training 8 minutes, and flexibility training for 7 minutes. They will receive a weekly check-in to discuss the exercises and progress with the QEP who will adjust the exercises based on tolerance. During the first session of each of the 12- weeks, a video about a health topic by an expert will be shown on Zoom so that they can think about it after the class and prepare questions for the discussion with the expert.

Their support person are invited to participate in this study. We assume that involving support persons in this study, including exercising together, can improve the health and quality of life of the patient and and their support person. If they or their support person do not have a tablet/laptop to join the class, this will be provided along with training on how to use them.

The control group will receive usual care and the option to receive the intervention after 12 weeks.

May 2024. We have added a single pre-post test group for patients who receive the geriatric assessment already in the older adults with cancer clinic. These participants will receive the 12 week virtual intervention and will not be randomized. They will be in the study for 12 weeks (no waitlist control period).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65+ years.
2. Diagnosed with lung, gastrointestinal (GI) , breast, Gynecologic or Genitourinary (GU) cancer or lymphoma who are referred for chemotherapy or immunotherapy and have not received > 4 weeks of systemic treatment.

4) Have a physician estimated life expectancy of >6 months. 5) Be physically inactive (no more than 90 min moderate to vigorous activity per week as per GLTEQ and do not currently meet the recommended physical activity volume of 90 min of aerobic exercise/week).

6) Able to speak and understand English. 7) Able to give informed consent. 8) Are considered safe to participate in the weekly classes as per their treating oncologist.

Eligible support persons are:

1. Identified by the older adult as their support person.
2. Aged 18 years and over.
3. Able to speak and understand English.
4. Able to give informed consent.

Exclusion Criteria:

1. Severe neuropsychiatric abnormalities (e.g., moderate-severe dementia) per the treating physician; and
2. Clinic visit with a geriatrician in the previous 12 months (they have already received part of the intervention).
3. Chest tube in-situ.

Exclusion criteria support person:

Not able to give informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasability of the study | 12 weeks
  What is the feasibility of implementation of the study? Feasibility will be measured by recruitment rate which will be the proportion of eligible patients and support persons who agree to enroll in the study, collected from our recruitment log) and measured in percentage with range 0-100. Feasibility of retention will be measured proportion of participants who complete the study data collection, collected from our study log), range 0-100.
  Feasibility of data outcome collection will be the percentage of patients who have complete data collection (collected from our study log), range 0-100.
  Feasibility of the study will be defined as recruitment of >60% of all eligible older adults; retention of >80% of the dyads; and 3) capture of outcome data of 80% or more.
Acceptability of the intervention and the study | 12 weeks
  What is the acceptability of the intervention and study? Acceptability will be measured by 1) adherence to the intervention and 2) satisfaction. Adherence to the intervention= 1) adherence to the geriatric assessment recommendations (collected through chart review) and expressed as percentage of recommendations received and implemented by the patient, range 0-100. 2) Adherence to online classes will be measured through the number of sessions missed as documented in the intervention log.
  A 5-item Likert scale satisfaction with the study scale ranging from very satisfied to very unsatisfied and satisfied and very Satisfied= satisified.
  Acceptability will be defined as 1) adherence to the intervention of >85% of participants adhering to at least 80% of the classes and recommendations; 2) satisfaction by 80% of participants.

SECONDARY OUTCOMES:
Effect intervention on Physical function | 12 weeks
  What are the preliminary estimate of the intervention on physical function? This will be measured with the Short Physical Performance Battery (SPPB). The Short Physical Performance Battery is a test battery comprising of a four-meter gait speed test, a balance test, and 5 timed chair stand tests. The total score ranges between 0-12, and a change of one point is considered the minimal clinically important difference (MCID).
Effect intervention on Grip strength | 12 weeks
  What are the preliminary estimates of the intervention on grip strength? Grip strength in kilos will be measured with a handheld dynamometer three times in the dominant hand (range 0-80 kg). The maximum score will be used, and the minimal clinically important difference (MCID) is 5 kg.
Effect intervention on Life space Mobility | 12 weeks
  What are the preliminary estimates of the intervention on Life Space Mobility? Life Space Mobility (LSM) will be measured with the University of Alabama Birmingham Study of Aging Life Space Assessment. The Life Space Mobility total score ranges from 0 (bed-bound) to 120 (daily independent out-of-town mobility). The minimal clinically important difference (MCID)is five points.
Effect intervention on Physical Activity | 12 weeks
  What are the preliminary estimates of the intervention on Physical Activity? Physical activity will be measured with the Godin Leisure time Exercise questionnaire. It asks how many times in the past seven days the participant has done vigorous, moderate, and light exercise for at least 15 min each time, and how much time the participant spent on the exercise, to calculate the total score. A score of 24+ indicates Active, 14 - 23 indicates Moderately Active, and <14 indicates inactive/sedentary
Effect intervention on number of self-reported Falls | 12 weeks
  What are the preliminary estimates of the intervention on the number of self-reported falls? Self-reported falls will be assessed weekly by a phone call by the RA as well as circumstances of the fall and will be scored as the total number of falls (ranging from 0- 200).
Effect of the intervention on Fatigue | 12 weeks
  What are the preliminary estimates of the intervention on fatigue? This will be measured with the Pittsburgh Fatigability questionnaire (PFS). The Pittsburgh Fatigability questionnaire measures both physical and mental fatigability. Participants rate their tiredness/exhaustion from 0 ("no fatigue") to 5 ("extreme fatigue") for how they expected or imagined they would feel after completing activities ranging in type and intensity (10 items). Continuous scores for each dimension can range from 0 to 50, with higher scores indicating higher fatigability and scores >25 will be used to indicate severe fatigability.
Effect of the intervention on Quality of life | 12 weeks
  What are the preliminary estimates of intervention on quality of life? This will be measured with the 12-item Short Form Survey (SF-12) . The 12 items are summarized in a physical subscale ranging from 0-100 and a mental health subscale ranging from 0-100.
Effect of the intervention on treatment toxicity | 12 weeks
  What are the effect of the intervention on Treatment toxicity ? This will be abstracted from the medical charts and treatment toxicity will be graded using the Common Terminology Criteria for Adverse Events version 5.0. Each toxicity is graded from 0-5. The number of toxicities grade 3-5 will be summed.
Effect of the intervention on unplanned healthcare utilization | 12 weeks
  What are the effect of the intervention on unplanned Emergency Department (ED) visits and/or hospitalization? This will be abstracted from the medical charts and summarized as the number of unplanned emergency department visits and number of unplanned hospitalizations. Both could range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Puts, RN PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jebanesan N, Alibhai SMH, Santa Mina D, Jones J, Legacy N, Freeman L, Smith A, Cobbing S, Vadali N, Lo S, Godhwani K, Nasiri F, Antonio M, Stephens D, Pitters E, Bennie F, Stephens A, Papadakos J, Cerullo L, Zjadewicz M, Jang R, Eng L, Krzyzanowska M, Matthew A, Durbano S, Mehta R, Menjak I, Emmenegger U, Sattar S, Sun V, Ladham K, Puts M. Supporting older adults with cancer and their support person through geriatric assessment and remote exercise and education: The SOAR study protocol. J Geriatr Oncol. 2025 Apr;16(3):102194. doi: 10.1016/j.jgo.2025.102194. Epub 2025 Feb 5. PMID 39909737